CLINICAL TRIAL: NCT07389200
Title: Application of Multimodal MRI-based Radiomics in Histological Grading and Prognostic Assessment of Breast Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Hao Xu (Other)
Responsible Party: Sponsor-Investigator, Hao Xu, Clinical Professor of Department of Radiology, Sichuan Cancer Hospital & Institute, Sichuan Cancer Hospital and Research Institute
Organization: Sichuan Cancer Hospital and Research Institute (Other)
Other Study IDs: SCCSMC-01-2024-119
Record Dates: First submitted 2026-01-10; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Breast Cancer With Low to Intermediate HER2 Expression
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 400 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast Cancer
  Interventions: Other: DCE-MRI

INTERVENTIONS:
Other: DCE-MRI — Patients at Hospital 1 underwent DCE-MRI using a 16-channel breast coil on a 3.0-T MRI scanner (Skyra, Siemens Healthcare, Erlangen, Germany) for the training and internal validation set. The external validation set comprised patients from Hospital 2 (GE Signa HDxt, equipped with a dedicated 7-channel phased-array breast coil) and Hospital 3 (Ingenia, Philips, Amsterdam, the Netherlands, also featuring a dedicated 7-channel phased-array breast coil)

SUMMARY:
In addition to TNM staging, the current management of breast cancer is based on conventional pathological features that categorize the disease into three molecular subtypes, each with significant prognostic implications in clinical practice: human epidermal growth factor receptor 2 (HER2)-positive, luminal (hormone receptor-positive and HER2-negative), and triple-negative breast cancers. The overexpression or amplification of HER2 is observed in 10-15% of breast cancer cases. This phenomenon often correlates with a more aggressive tumor behavior while also demonstrating an increased responsiveness to HER2-targeted therapies. However, the use of highly effective anti-HER2 drugs can significantly enhance the survival outcomes of these patients. Additionally, the expression status of HER2 is critical in determining the necessity for targeted therapy. Therefore, preoperative assessment of HER2 expression status has important therapeutic implications. Currently, clinical methods for assessing HER2 status in breast cancer before surgery include immunohistochemistry (IHC) tests and fluorescence in situ hybridization (FISH) measurements performed on core-needle biopsy specimens. However, these biopsy sampling techniques have inherent limitations, including sampling bias and an inability to fully represent intratumor heterogeneity. Additionally, the biopsy procedure can be uncomfortable and carries certain risks for patients. Tumour heterogeneity generally refers to the variations in angiogenesis, metabolism, gene expression, and other biological characteristics among tumors. Intratumoral heterogeneity (ITH) can manifest as signal differences in radiological images at the macro level. Investigators hypothesized that significant differences in biological characteristics and behavior exist between HER2-positive (HER2+) and HER2-negative (HER2 -) breast cancers, allowing for the distinction of these two types of tumours by identifying specific imaging features that reflect ITH.

Dynamic contrast-enhanced MRI (DCE-MRI) is an effective imaging modality that provides temporal information regarding the dynamics of contrast agents in suspicious lesions while maintaining acceptable spatial resolution. It is particularly sensitive in detecting breast cancer lesions, especially those in dense breast tissue. DCE-MRI can indirectly reflect abnormal tumor vascular proliferation through the hemodynamic characteristics of the lesions. Radiomics is an emerging technology that involves extracting quantitative and reproducible features from medical images using high-throughput, sophisticated modalities that are often challenging to identify or quantify visually. These features, which may be linked to specific diseases, are analyzed using statistical or machine learning (ML) algorithms to create predictive models for tumor diagnosis, grading, efficacy evaluation, and prognosis prediction. ML has two important advantages over traditional statistical models. The goal is to reduce decision time during diagnosis and generally achieve greater diagnostic accuracy. As demonstrated in breast cancer diagnosis, ML can significantly improve cancer risk prediction by identifying complex patterns in large amounts of clinical data. Despite the great potential of ML, it still faces several obstacles in its clinical application. A major challenge is a lack of interpretability-many ML models operate like "black boxes", making it difficult for clinicians to understand and trust their decision-making processes. Furthermore, the performance of the model depends heavily on the quality and representativeness of the training data. ML methods often require larger data sets than traditional clinical studies.

Thus, this study aimed to develop a radiomics-based ML model that could predict the HER2 status of breast cancers in a non-invasive manner using DCE-MRI images. Additionally, the Shapley Additive Explanation (SHAP) algorithm was employed to analyze the contribution of the variables included in the model, providing valuable insights for formulating more accurate preoperative treatment plans for patients with breast cancers.

ELIGIBILITY:
Inclusion Criteria:

* Histopathological diagnosis of breast cancer by surgical or biopsy pathology;
* Availability of DCE-MRI within two weeks before surgery
* No prior treatment before baseline DCE-MRI examination.

Exclusion Criteria:

* Less than 5 mm of long diameter of the lesion
* Severe motion artifacts
* Missing or incomplete essential data
* Anti-tumor treatment before MRI

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 368 female patients diagnosed with breast cancer from three hospitals between August 2017 and December 2021 were consecutively recruited in this study
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2028-01-01 (Estimated); Primary Completion 2029-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Patients with pathologically confirmed breast cancer who underwent DCE-MRI were included. Radiomic features were extracted, and seven machine learning algorithms were utilized to construct predictive model.The AUC served as the evaluation metric | From enrollment to the end of treatment at 8 weeks
  The AUC served as the primary evaluation metric for identifying the optimal model. A comprehensive model evaluation was conducted, which included AUC, accuracy, sensitivity, specificity
F1 score | From enrollment to the end of treatment at 8 weeks
  F1 score, with validation on an independent cohort.

SECONDARY OUTCOMES:
histopathological diagnosis of breast cancer by surgical or biopsy pathology | From enrollment to the end of treatment at 8 weeks

OTHER OUTCOMES:
To investigate the correlation between biological and radiomics features, we compared the diferences in radiomics features selected by SHAP between diferent Ki67 index and hormone receptor status | From enrollment to the end of treatment at 8 weeks

IPD SHARING:
Plan to Share IPD: No